CLINICAL TRIAL: NCT05194241
Title: Examining the Efficacy of a Single Session Mindfulness Oriented Recovery Enhancement Intervention: One MORE
Brief Title: One MORE for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 00146987
Record Dates: First submitted 2021-11-16; First posted 2022-01-18 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain
Keywords: Mindfulness
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One MORE (Experimental)
  Interventions: Behavioral: One MORE
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: One MORE — One MORE is a 2-hour adaptation of the manualized MORE program and will be divided into four, 30-minute segments. In the first segment, participants will be introduced to mindfulness and guided though a body scan practice, which directs participants to systematically shift attention from one part of the body to the next. Mindful pain management will be the focus of the second segment and participants will be guided through a mindfulness of pain practice in which they will learn to deconstruct pain into sensory, emotional, cognitive, and behavioral components. The third segment will focus on managing the negative thoughts and emotion that can amplify pain with mindful reappraisal, and the fourth segment will focus on increasing the positive emotions that can attenuate pain with mindful savoring.
  Arms: One MORE

SUMMARY:
This study will be a single-site, two-arm randomized controlled trial conducted among chronic pain patients. Chronic pain patients will be randomized by a computer-generated randomization schedule with simple random allocation (1:1) to either One MORE or a wait-list control condition (WLC). One MORE will be delivered individually via a HIPAA compliant virtual meeting platform.

ELIGIBILITY:
Inclusion Criteria:

* men/women ≥18 years of age
* current chronic pain diagnosis
* reporting pain ≥3 on 0-10 scale

Exclusion Criteria:

* unstable illness judged by clinician to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Pain Catastrophizing | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in pain catastrophizing from baseline through 3-month follow-up will be assessed with the Pain Catastrophizing Scale. Scores range from 0 to 52, with higher scores reflecting greater pain catastrophizing.

SECONDARY OUTCOMES:
Pain Intensity | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in pain intensity from baseline through 3-month follow-up will be assessed with the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain intensity.
Pain Interference | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in pain interference from baseline through 3-month follow-up will be assessed with the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 20, with higher scores reflecting greater pain interference.

OTHER OUTCOMES:
Physical Function | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in physical function from baseline through 3-month follow-up will be assessed with the PROMIS Physical Functioning Short Form. Scores range from 6 to 30, with higher scores reflecting greater physical function.
Sleep | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in sleep from baseline through 3-month follow-up will be assessed with the PROMIS Sleep Disturbance Short Form. Scores range from 6 to 30, with higher scores reflecting worse sleep.
Depression | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in depression from baseline through 3-month follow-up will be assessed with the Patient Health Questionnaire-2. Scores range from 0 to 6, with higher scores reflecting greater depression.
Anxiety | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in anxiety from baseline through 3-month follow-up will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.
Prescription Pain Medication Misuse | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in prescription pain medication misuse from baseline through 3-month follow-up will be assessed with the PROMIS Prescription Pain Medication Misuse Short Form. Scores range from 7 to 35, with higher scores reflecting greater medication misuse.
Trait Mindfulness | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in trait mindfulness from baseline through 3-month follow-up will be assessed with the Toronto Mindfulness Scale - Trait Version. Scores range from 0 to 52, with higher scores reflecting greater trait mindfulness.
Trait Self-Transcendence | Will be completed at baseline, week 2, and 1, 2, and 3 months after baseline.
  Change in trait self-transcendence from baseline through 3-month follow-up will be assessed with the Nondual Awareness Dimensional Assessment - Trait Version. Scores range from 0 to 52, with higher scores reflecting greater trait self-transcendence.
Acute Pain | Will be completed immediately before and after the 2-hour, One MORE intervention.
  Change in acute pain will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain.
Decentering | Will be completed immediately before and after the 2-hour, One MORE intervention.
  Change in decentering will be measured with the state version of the Metacognitive Processes of Decentering scale. Scores range from 0 to 10, with higher scores reflecting greater decentering.
Self-Transcendent State | Will be completed immediately before and after the 2-hour, One MORE intervention.
  Change in self-transcendent state will be measured with the Nondual Awareness Dimensional Assessment - State Version. Scores range from 0 to 10, with higher scores reflecting greater self-transcendence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hanley AW, Lingard A, Garland EL. A Single-Session, 2-Hour Version of Mindfulness-Oriented Recovery Enhancement (One MORE) Improves Chronic Pain Patients' Pain-Related Outcomes Through 3-Month Follow-Up in a Randomized Controlled Trial. J Integr Complement Med. 2024 Sep;30(9):869-877. doi: 10.1089/jicm.2023.0501. Epub 2024 Apr 8. PMID 38588552